CLINICAL TRIAL: NCT01653210
Title: Development of an Advisory System for Glycemic Control During the Menstrual Cycle in Patient With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: LifeScan (Industry)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Other Study IDs: 16272
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin Pump; Continuous Glucose Monitor; Premenopausal women
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At each follow-up visit #3-13, blood will be taken to sample estradiol, progesterone, luteinizing hormone (LH), follicle-stimulating hormone (FSH), total testosterone and sex-hormone binding globulin (SHBG). At the end of study visit #14, a hemoglobin A1c will be measured.
Oversight: Data Monitoring Committee: No

SUMMARY:
This overall research goal will be to develop a mobile-based module to improve glycemic control during the menstrual cycle in women with Type 1 diabetes mellitus (T1DM). This module will run on an Android Operating System (OS) and will be available as: (i) a stand-alone application and (ii) an important additional component to a larger system, the Diabetes Assistant (DiAs) - a mobile-based medical platform for diabetes applications. This proposal aims to build one such application or module targeting the improvement of diabetes control in younger women who experience glucose variation related to their menstrual cycle.

DETAILED DESCRIPTION:
The purpose of this particular protocol is to study the underlying glycemic variability across the menstrual cycle in women with T1DM. A subset of premenopausal women with T1DM experience loss of glucose control during the latter half of the cycle (the luteal phase). Clinical trials are sparse and tools are limited to focus on this aspect of diabetes care which is highly relevant in affected individuals. To obtain data to initialize this mobile-based module, we will enroll premenopausal women for approximately three-month outpatient study designed to characterize at least three complete menstrual cycles. These subjects will wear continuous glucose monitors (CGMs), record self-monitored blood glucoses (SMBGs) and utilize an insulin pump to capture insulin dosing. In-home ovulation kits will be used to determine relevant days for sex-steroid blood measurements to define menstrual cycle phases. Finally, structured at-home meals will be provided during different phases of the menstrual cycle for insulin action parameters assessments.

The software module will be developed in parallel with the data collection from study subjects. The software module will not be used with the patients in this study as it is not in existence as would be developed in parallel. The goal of the module functionality will be to 1) assist patients and providers in the identification and management of glycemic variability surrounding the menstrual cycle and 2) add value to and become an integral module within the artificial pancreas.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women with menstrual cycles that occur approximately every 20-40 days.
2. T1DM (as defined by the American Diabetes Association criteria or judgment of a physician) for at least 2 years prior to the enrollment in the study
3. Age ≥18 y.o. and ≤55 y.o.
4. Use of an insulin pump to treat their diabetes for at least 6 months.
5. Has an identified healthcare provider who can provide advice about diabetes care.
6. Actively using a current insulin pump with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor.
7. Willingness to do additional fingersticks when requested such as when CGM alarms at low or high end (<70 mg/dl or >300 mg/dl),
8. Willingness to come to Center for Diabetes Technology for study visits.
9. Willingness to avoid consumption of acetaminophen-containing products for the duration of the study.
10. Demonstration of proper mental status and cognition for completion of the study.
11. Hemoglobin A1c 5-10%

Exclusion Criteria:

1. Pregnant or intending to get pregnant during study
2. Active enrollment in another clinical trial
3. Medical requirement for acetaminophen-containing products during the study period for more than 1 week
4. Use of medication or intervention that significantly alters the menstrual cycle such as oral contraceptives, depoprovera, or intrauterine device (IUD).
5. Medical condition that would make operating a CGM or insulin pump difficult (e.g. blindness, severe arthritis, extensive scar tissue at sites where devices are inserted)
6. Anticipated need for Magnetic resonance imaging (MRI)/Magnetic resonance angiography (MRA) during the study. Unplanned MRI/MRA requiring temporary interruption of CGM use would be allowed.
7. Use of prednisone for more than 10 days during the study.
8. Uncontrolled thyroid disease
9. Clinical diagnosis of polycystic ovarian syndrome requiring treatment.
10. Significant elevation in liver function tests (e.g. >2-3 times normal), known infectious hepatitis or HIV.
11. History of a systemic deep tissue infection with methicillin-resistant staph aureus or Candida albicans
12. Known bleeding diathesis or dyscrasia
13. Active renal dialysis
14. Individuals with cognitive impairment that prevents understanding either consent form or intervention content
15. Psychiatric disorders that would interfere with study tasks (e.g., substance abuse)-self reported

List any restrictions on use of other drugs or treatments.

1. Acetaminophen with the use of the CGM.
2. Use of medication or intervention that significantly alters the menstrual cycle such as oral contraceptives, depoprovera, or IUD.
3. Anticipate need for MRI/MRA during the study. Unplanned MRI/MRA requiring temporary interruption of CGM use would be allowed.
4. Use of prednisone for more than 10 days during the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fifteen premenopausal women with menstrual cycles, 18-55 years of age, who have been diagnosed as type 1 diabetic for at least 2 years. Actively using a current insulin pump for the past 6 months with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor. Use of medication or intervention that significantly alters the menstrual cycle such as oral contraceptives, depoprovera, or intrauterine device (IUD)is prohibited.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue A. Brown, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Direct request of Principal Investigator.

RESULTS

PARTICIPANT FLOW:
Groups:
- Female T1DM: Premenopausal women with menstrual cycles, 18-55 years of age, who have been diagnosed as type 1 diabetic for at least 2 years. Actively using a current insulin pump for the past 6 months with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor. Use of medication or intervention that significantly alters the menstrual cycle such as oral contraceptives, depoprovera, or intrauterine device (IUD)is prohibited.
Period: Overall Study
Arm/Group | Female T1DM
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Female T1DM
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: High Blood Glucose Index (HBGI)
Description: Measure of Hyperglycemic Risk based on frequency and severity of hyperglycemic events.
  HBGI < 4.5 is associated with lower risk of hyperglycemia, 4.5 < HBGI < 9 is associated with a moderate risk of hyperglycemia and HBGI > 9 is associated with high risk of hyperglycemia.
  Our primary outcome measure is hyperglycemia risk during the luteal phase of the menstrual cycle. The primary hypothesis is there is an increased hyperglycemia risk during the luteal phase when compared to the follicular phase. Subjects will be compared to themselves across the three menstrual cycles captured. Hyperglycemia will be primarily assessed by high blood glucose index which was assessed over 3 menstrual cycles at specific time points in the cycle.
Time Frame: Three menstrual cycles (average length of one cycle was 28.7 days)
Measure: Mean (Standard Error); unit: index score
Arm/Group | Female T1DM
Number analyzed (Participants) | 12
index score
  Early Follicular | 6.87 (0.88)
  Mid-Late Follicular | 8.05 (1.08)
  Peri-Ovulation | 7.92 (1.13)
  Early Luteal | 9.00 (1.25)
  Mid Luteal | 8.02 (0.99)
  Late Luteal | 7.50 (0.91)
Statistical Analysis 1: Comparison: Female T1DM; Test type: Superiority or Other; p = 0.023, ANOVA

2. Secondary Outcome: Glycemic Changes During Luteal Phase
Description: Changes in estrogen and progesterone will be primary drivers of hyperglycemia risk during the luteal phase. These data will be analyzed as continuous variables.
Time Frame: Three Menstrual Cycles
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Female T1DM
Number analyzed (Participants) | 12
pg/mL
  Estradiol: Early Follicular | 41.34 (3.7)
  Estradiol: Mid-late Follicular | 91.79 (13.77)
  Estradiol: Periovulation | 225.06 (43.69)
  Estradiol: Mid-Luteal | 213.33 (23.15)
  Estradiol: Late Luteal | 143.81 (15.19)

ADVERSE EVENTS:
Groups:
- Female T1DM: Twelve premenopausal women with menstrual cycles, 18-55 years of age, who have been diagnosed as type 1 diabetic for at least 2 years. Actively using a current insulin pump for the past 6 months with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor. Use of medication or intervention that significantly alters the menstrual cycle such as oral contraceptives, depoprovera, or intrauterine device (IUD)is prohibited.
Arm/Group | Female T1DM
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes